CLINICAL TRIAL: NCT01095965
Title: Implementation and Evaluation of a Nutrition Education Programme for Adults With Type 2 Diabetes Mellitus in a Resource Poor Setting of the Moretele Sub-District, North West Province, South Africa
Brief Title: Nutrition Education Intervention in Adults With Type 2 Diabetes Mellitus in a Resource Poor Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pretoria (Other)
Collaborators: South African Sugar Association (Unknown); Nestlè Nutrition Institute Africa (Other)
Responsible Party: Principal Investigator, Jane Muchiri, PhD Student, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MuchiriUP; DOH-27-0310-3070 (Other: South Africa Department of Health)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type II [Non-insulin Dependent Type] [NIDDM Type] Uncontrolled
Keywords: Nutrition education intervention; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle education (Experimental): Nutrition education comprised of 4 components: Curriculum (8 weeks), follow-up meetings (4 monthly plus 2-bimonthly), education materials for use at home and vegetable gardening demonstrations.
  Interventions: Behavioral: Nutrition education

INTERVENTIONS:
Behavioral: Nutrition education — Group education on a bi-weekly basis for eight weeks plus written education materials, followed by monthly group problem solving meetings till one year.

SUMMARY:
The purpose of this study is to implement a nutrition education programme that was developed for type 2 diabetic adults in a resource poor setting and to evaluate the programme's effectiveness on health outcomes

A randomized controlled clinical trial study design will be used. One group (experimental group) will receive the nutrition education while the other group (control group) will receive the usual care.

Setting: Two Community health centres in Moretele Health Sub-District, North West Province, South, Africa

Effectiveness of the nutrition education will be evaluated for the following outcomes:

* clinical

  * blood sugar control based on HbA1c levels (primary outcome)
  * lipid profile (total cholesterol, low density cholesterol, high density cholesterol and triglycerides)
  * blood pressure
  * body mass index
* dietary intake
* others -diabetes knowledge, attitudes towards diabetes

Outcome measurements- at six and 12 months, this will be compared with the baseline data.

Hypotheses:

* the experimental group will have a significantly lower HbA1c compared to the control group
* the experimental group will have significantly better outcomes for dietary intake, blood lipid profile, blood pressure, body mass index, diabetes knowledge and attitudes towards diabetes and its treatment.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (DM) is a global health challenge. Low-income individuals are among those observed to have poorer long term outcomes of diabetes management and to spend a higher proportion of their income on diabetes care. Therefore, diabetic individuals from resource poor settings require special attention and effective management strategies to assist them improve their health outcomes. Patient self-management education, including nutrition education is a feasible strategy in resource poor settings.

The nutrition education programme in this study is based on the target group assessed needs, as tailored education is shown to be more effective in improving health outcomes.

The experimental group will receive nutrition education in group format on a weekly basis for eight weeks, this will include a vegetable gardening component offered in collaboration with the Department of Agriculture. In addition written education materials will be provided (pamphlet and wall/fridge flyer). A follow-up intervention on a monthly basis will follow the group education.This is to revise the learnt content and for group problem solving activities. The control control group will receive usual care plus the written education materials.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* 40 to 70 years
* At least one year living with diabetes
* Blood sugar levels of 10mmol/L or above in at least two occasions in the last six months and consequent HbA1c levels of ≥8mmol/L
* Regular attendance of diabetic clinic

Exclusion Criteria:

* On insulin therapy
* Pregnant
* Full time employment
* Plans to move from study area during the study period

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
HbA1c as a measure of glycemic control | 12 months
  % change from baseline, 6 months and 12 months

SECONDARY OUTCOMES:
Dietary intake | 12 months
  Contribution of macronutrients to total energy intake, intake of fibre, intake of micronutrients, portion sizes, intake of fruits and vegetables, change from baseline, 6 months and 12 months
Lipid profile | 12 months
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, tryglycerides, changes from baseline, 6 months and 12 months
Blood pressure | 12 months
  Change in blood pressure from baseline, 6 months and 12 months
Diabetes knowledge | 12 months
  Change in knowledge levels from the baseline, 6 months and 12 months
Attitudes toward diabetes and its treatment | 12 months
  Change in attitudes from baseline, 6 months and 12 months
Body mass index | 12 months
  Change from baseline, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jane W Muchiri, PhD, Principal Investigator — University of Pretoria; Paul Rheeder, PhD, Study Chair — University of Pretoria
Locations (1):
- Moretele Health Sub-District, Hammanskraal, North West, South Africa